CLINICAL TRIAL: NCT07174947
Title: SSRI Antidepressant Fluoxetine Improving Immunotherapy Efficacy in Advanced Hepatobiliary Malignancy Patients With Depression and Anxiety: A Randomized Controlled Clinical Trial
Brief Title: SSRI Antidepressant Fluoxetine Improving Immunotherapy Efficacy in Advanced Hepatobiliary Malignancy Patients With Depression and Anxiety
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Gang Chen, MD, M.D., Ph.D., First Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSRI
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Hepatobiliary Malignancy; Fluoxetine; Anxiety Disorders; Depression Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Fluoxetine; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): 1. Standard treatment plan For patients with hepatocellular carcinoma, the first-line treatment regimen containing PD-1 inhibitors /PD-L1 inhibitors is adopted: 1) Toripalimab + bevacizumab 2) Tislelizumab 3) Nivolumab + ipilimumab For patients with cholangiocarcinoma, the combination of PD-1 inhibitors /PD-L1 inhibitors and gemcitabine + cisplatin/oxaliplatin (such as pembrolizumab +GEM -CDDP or durvalumab +GEM -CDDP) is adopted. 2. Fluoxetine: Maintain at 20mg per day, orally, until disease progression or intolerance. 3. The use of antiemetic, analgesic and other symptomatic treatment drugs is allowed, and all concurrent medication situations should be recorded.
  Interventions: Drug: Fluoxetine (drug)
- Control Group (Placebo Comparator): 1. Standard treatment plan
  For patients with hepatocellular carcinoma, the first-line treatment regimen containing PD-1 inhibitors /PD-L1 inhibitors is adopted:
  1. Toripalimab + bevacizumab
  2. Tislelizumab
  3. Nivolumab + ipilimumab For patients with cholangiocarcinoma, the combination of PD-1 inhibitors /PD-L1 inhibitors and gemcitabine + cisplatin/oxaliplatin (such as pembrolizumab +GEM -CDDP or durvalumab +GEM -CDDP) is adopted.
  2. Placebo: Take 1 placebo tablet per day for maintenance, orally.
  3. The use of antiemetic, analgesic and other symptomatic treatment drugs is allowed, and all concurrent medication situations should be recorded.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine (drug) — Fluoxetine: Maintain at 20mg per day, orally, until disease progression or intolerance
  Arms: Experimental Group
Drug: Placebo — Placebo: 1 placebo tablet per day for maintenance, orally.
  Arms: Control Group

SUMMARY:
Advanced liver and gallbladder malignancies (including liver cancer, cholangiocarcinoma and gallbladder cancer) are a type of disease that is difficult to treat, and most patients have a short survival period. In recent years, immunotherapy (such as PD-1/PD-L1 inhibitors) has brought new hope to these patients, but still only a small number of patients can benefit.

Research has found that approximately 40% of patients with liver and gallbladder tumors have symptoms of depression and anxiety, which not only affect their quality of life but may also reduce the therapeutic effect by influencing immune function. Fluoxetine is a commonly used antidepressant. The latest research shows that in addition to improving mood, it may also enhance the anti-tumor effect of immunotherapy. This study aims to explore whether fluoxetine combined with immunotherapy can better control tumors than immunotherapy alone, prolong the survival period of patients, and at the same time improve the depressive and anxious symptoms and quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 80 years old, both male and female are acceptable.
* The histopathological/cytological diagnosis is hepatocellular carcinoma or cholangiocarcinoma. Hepatocellular carcinoma can be diagnosed by imaging.
* Patients with metastatic advanced or locally advanced liver and gallbladder malignancies;
* No treatment has been received and a first-line treatment regimen including PD-1 inhibitors /PD-L1 inhibitors is planned to be carried out;
* Patients with a PHQ-9 score of ≥10 or a GAD-7 score of ≥8, that is, those with positive screening for depression or anxiety;
* At least one lesion measurable by CT or MRI (with a maximum diameter of ≥0.5cm);
* ECOG: 0-2;
* Child-Pugh score ≤7 points;
* The expected survival period is ≥12 weeks.
* Baseline blood cell count tests and blood biochemistry must meet the following standards:1) White blood cell count ≥3.0×10^9/L; Hemoglobin ≥90 g/L;2) Absolute neutrophil count ≥1.5×10^9/L;3) Platelet count ≥100×10^9/L;4) Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of the normal upper limit (ULN);5) Total bilirubin ≤ twice ULN;6) Serum creatinine ≤ 1.5 times ULN; Albumin ≥30 g/L;
* The subjects voluntarily joined this study, signed the informed consent form, had good compliance and cooperated with the follow-up.

Exclusion Criteria:

* Those with uncorrectable coagulation dysfunction and a distinct bleeding tendency;
* Patients who currently have unstable or active ulcers or gastrointestinal bleeding;
* Severe functional insufficiency of vital organs, such as severe cardiopulmonary insufficiency, etc;
* Patients with hepatic encephalopathy or intractable ascites requiring treatment;
* A history of mental disorders such as bipolar disorder, schizophrenia, and active suicidal ideation;
* Patients with active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (active is defined as a viral load > 20,000 IU/mL), or those who are positive for HBV or HCV and refuse to receive standardized antiviral treatment;
* Unable to swallow oral medication;
* Patients allergic to fluoxetine;
* Currently using drugs that may have serious interactions with fluoxetine;
* The researchers assessed that the patient was unable or unwilling to comply with the requirements of the research protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by mRECIST (%) | at 4-12 weeks after treatment initiation
  Proportion of participants achieving complete response (CR) or partial response (PR) based on mRECIST criteria, measured on contrast-enhanced CT/MRI at 4-12 weeks after treatment initiation.

SECONDARY OUTCOMES:
Overall Survival (OS) (months) | 5 years
  Time from treatment initiation to death from any cause.
Progression-Free Survival (PFS) (months) | 5 years
  Time from treatment initiation to radiologically confirmed disease progression (mRECIST) or death from any cause, whichever occurs first.
status of anxiety and depression | 5 years
  measured by psychologist using GAD-7 and PHQ-9, more than 10 points in either of the charts would be marked as positive
Quality of Life Score (EORTC QLQ-C30, 0-100 scale) | 5 years
  Health-related quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30). Scores for global health status/QoL, functional scales, and symptom scales will be calculated according to the EORTC scoring manual, with higher scores indicating better functioning for functional scales and worse symptoms for symptom scales.

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The individual participant data (IPD) that underlie the results reported in this article will be made available beginning 6 months after publication and ending 36 months after publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for use in achieving the aims of a specified research project. Proposals should be directed to corresponding author's email. To gain access, data requesters will need to sign a data access agreement.